CLINICAL TRIAL: NCT04531124
Title: Cardiovascular and Renal Outcomes of Integrated Management of Blood Pressure and Other Cardiometabolic Risks in Hypertensives：a Multicenter Prospective Cohort Study （UPDATE-cohort）
Brief Title: Cardiovascular and Renal Outcomes of Integrated Management of Blood Pressure and Other Cardiometabolic Risks in Hypertensives
Status: Not yet recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Yong Li, Professor, MD, PhD, Huashan Hospital
Other Study IDs: Huashan cardiology
Record Dates: First submitted 2020-08-15; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Cardiovascular Risk Factor; Hypertension; Renal Disease
MeSH Terms: conditions — Hypertension; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group without an integrated management
- observational group with an integrated management
  Interventions: Other: integrated management

INTERVENTIONS:
Other: integrated management — establish an integrated management on cardio-metabolic risk factors including hypertension by updating and upgrading the daily practice of practitioners and screening patients
  Groups: observational group with an integrated management

SUMMARY:
this clinical trial is designed to study the cardiovascular and renal outcomes of hypertensives after an integrated management of blood pressure and other cardiometabolic risks. it is a multicenter prospective cohort study.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients from departments of Cardiology, Endocrinology, Nephrology, Neurology, Geriatrics or General Internal Medicine.
2. Diagnosed as hypertension. Diagnostic criteria: 1)The office BP measured at the day of visit and at least one time before that day were above the cut-off values ( ≥140 mmHg SBP and/or ≥90 mmHg DBP); 2)for patients with normal BP at the day of visit, they should have already been given pre-treatment with antihypertensive drugs ≥ 2 weeks.
3. Voluntary participation.

Exclusion Criteria:

1. Patients aged< 18 years old.
2. Patients without a definite diagnosis of hypertension(for instance, if the patient has been taking antihypertensive drugs irregularly, it is difficult to confirm the diagnosis of hypertension).
3. Patients with a definite diagnosis of secondary hypertension.
4. Patients are diagnosed dyslipidemia with clear cause, such as nephrotic syndrome, severe hypothyroidism, terminal stage of malignancy, etc.
5. Patients are diagnosed end-stage renal disease, hemodialysis, and peritoneal dialysis patients.
6. Patients diagnosed with mental abnormalities who are unable to complete the questionnaire.
7. Patients have once participated in this research during this study cycle(to avoid repeated participation).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatients with hypertension in different levels of hospitals in Shanghai, China
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
complex outcome | follow-up 1 year
  number of participants with 3P-MACE events(cardiovascular deaths, non-fatal myocardial infarction, non-fatal stroke)
coronary angioplasty | follow-up 1 year
  number of participants with coronary angioplasty
acute renal failure | follow-up 1 year
  number of participants with acute renal failure(eGFR decreases by 50% or <15ml/min/1.73m2, dialysis or renal death)
acute heart failure | follow-up 1 year
  number of participants with acute heart failure(non-scheduled hospitalizations due to heart failure or required intravenous medication)

CONTACTS AND LOCATIONS:
Locations (1):
- HuashanH, Shanghai, Shanghai Municipality, China